CLINICAL TRIAL: NCT06078553
Title: Multicenter, Multinational, Natural History Study in Participants With Congenital Myasthenic Syndromes Due to Mutations in DOK7, MUSK, AGRN, or LRP4
Brief Title: A Natural History Study in Participants With Congenital Myasthenic Syndromes (CMS) Due to Mutations in DOK7, MUSK, AGRN, or LRP4
Status: Recruiting | Type: Observational
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Other Study IDs: ARGX-119-NIS-2301
Record Dates: First submitted 2023-09-08; First posted 2023-10-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Congenital Myasthenic Syndrome
MeSH Terms: conditions — Myasthenic Syndromes, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants will attend up to 4 study visits to collect clinical assessments. The assessments will evaluate participants' symptoms and quality of life to understand disease activity in patients with CMS due to mutations in DOK7, MUSK, AGRN, or LRP4.

ELIGIBILITY:
Inclusion Criteria:

* Can understand the requirements of the study and can provide written informed consent/assent, and willingness and ability to comply with the study protocol procedures
* Is male or female and aged ≥2 years at the time of providing informed consent/assent
* Has a diagnosis of CMS due to biallelic pathogenic mutations in DOK7 or any pathogenic mutations in MUSK, AGRN, or LRP4
* Has a total Quantitative Myasthenia Gravis (QMG) score of ≥3 (applies only to participants aged ≥6 years)
* For participants taking oral beta agonists (eg, albuterol, salbutamol, ephedrine), participant must have been receiving the medication for ≥3 months before screening/baseline

Exclusion Criteria:

* Known medical condition that would interfere with an accurate assessment of CMS, in the investigator's opinion
* Is currently participating in any interventional clinical study with a study drug at the time of providing informed consent/assent
* Diagnosis of CMS due to mutation of any gene other than DOK7, MUSK, AGRN, or LRP4

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with CMS due to mutations in DOK7, MUSK, AGRN, or LRP4 receiving standard of care at their treating physician
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Summary statistics of retrospective and prospective collection of data on diagnosis. | Up to 12 months
Summary statistics of retrospective and prospective collection of data on health care utilization. | Up to 12 months
Summary statistics of retrospective and prospective collection of data on medications. | Up to 12 months
Summary statistics of retrospective and prospective collection of data on change in health status related to CMS | Up to 12 months

SECONDARY OUTCOMES:
Change from baseline for QMG total score, each component score, and raw values | Up to 12 months
  The Quantitative Myasthenia Gravis (QMG) consists of 13 items that assess ocular, bulbar, and limb function. Six of the 13 items are timed endurance tests measured in seconds. Each item has a possible score from 0 to 3, with 3 being the most severe. The total possible score is 39, with higher scores indicating more severe impairments.
Change from baseline for MG-ADL total score | Up to 12 months
  The Myasthenia Gravis Activities of Daily Living (MG-ADL) is an 8-item scale that assesses MG symptoms and their effects on daily activities. The 8 items are rated by the participant on a scale of 0 to 3. The total score can range from 0 to 24, with higher total scores indicating more impairment.
Change from baseline for PROMIS-GHS | Up to 12 months
  The Patient-Reported Outcomes Measurement Information System Global Health Scale (PROMIS-GHS) is a quality-of-life questionnaire that comprises questions on overall physical health, physical function, pain, and fatigue (GPH); and quality of life, mental health, satisfaction with social activities, and emotional problems (GMH). The participant marks their response on a 5-point Likert scale, with lower scores indicating poorer health
Change from baseline for PROMIS-DFL | Up to 12 months
  The Patient-Reported Outcomes Measurement Information System Dyspnea Functional Limitations (PROMIS-DFL) is a questionnaire that evaluates the impact of dyspnea on the ability to perform daily activities within the last 7 days. The participant marks their response on a 4-point scale (0 to 3), with lower values indicating less functional impairment.
Change from baseline for EQ-5D-5L | Up to 12 months
  The EQ-5D-5L questionnaire is a standardized test recognized by many health authorities as a generic measure of health status for clinical and economic appraisal. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Participants mark their health status from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Change from baseline for 3TUG | Up to 12 months
  The Triple Timed Up and Go (3TUG) is an objective measure of mobility requiring 3 repetitions (laps) to assess lower extremity weakness and fatigability.
Change from baseline for Neuro-QoL Fatigue score | Up to 12 months
  The Quality of Life in Neurological Disorders (Neuro-QoL) Fatigue questionnaire will be completed by participants aged ≥18 years. The Neuro-QoL Pediatric Fatigue questionnaire will be completed by pediatric participants aged ≥12 to <18 years. Participants aged <8 years will be evaluated using the proxy version of the questionnaire.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (3):
  - UC Davis Health - UC Davis Health Midtown Ambulatory Care Center, Sacramento, California
  - Ann and Robert H Lurie Children's Hospital of Chicago - Main Hospital, Chicago, Illinois
  - Hospital Sisters Health System (HSHS) - St Elizabeth's Hospital, O'Fallon, Illinois
- Medical University of Vienna, Vienna, Austria
- The Ottawa Hospital - Civic Campus, Ottawa, Canada
- France (5):
  - CHU Bordeaux - Groupe Hospitalier Pellegrin - Neurology, Bordeaux
  - Hospices Civils de Lyon (HCL) - Hopital Pierre Wertheimer - Neurology, Bron
  - CHU Lille Hopital Salengro - Neurology, Lille
  - CHU Timone, Marseille
  - Assistance Publique Hopitaux de Paris - Hopital Pitie-Salpetriere, Paris
- Universitaetsklinikum Essen (AoR), Essen, Germany
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Centrum Medyczne Neurologia Slaska - Neurology, Katowice, Poland
- Spain (3):
  - Hospital Sant Joan de Deu - Pediatric Neurology, Esplugues de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - Ulster Hospital, Dundonald
  - Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital, Oxford